CLINICAL TRIAL: NCT02462720
Title: Multicenter Study to Evaluate Pain Following Treatment of Varicose Vein With Varithena® Compared to Radiofrequency Ablation
Brief Title: COMFORT: A Multicenter, Open-label, Randomized, Crossover Study
Acronym: COMFORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VAP.VV018
Record Dates: First submitted 2015-05-20; First posted 2015-06-04 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Polidocanol; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varithena®, then Radiofrequency Ablation (Experimental): Varithena (polidocanol injectable foam) supplied as polidocanol solution 180 mg/18 mL (10 mg/mL) to be activated before use. Once activated, Varithena is a white injectable foam delivering a 1% polidocanol solution. Each milliliter of Varithena injectable foam contains 1.3 mg of polidocanol. Up to 5 mL per injection or 15 mL per treatment session could be used. This was followed by RFA treatment.
  Interventions: Drug: Varithena®; Device: Radiofrequency ablation
- Radiofrequency ablation then Varithena (Active Comparator): RFA procedures were conducted in accordance with the physician's standard of care and according to the manufacturer's instructions for use. This was followed by treatment with Varithena.
  Interventions: Drug: Varithena®; Device: Radiofrequency ablation

INTERVENTIONS:
Drug: Varithena® — Varithena® treatment in accordance with full prescribing information and instructions for use
  Other Names: Polidocanol Solution, 180 mg/18 mL (10 mg/mL)
Device: Radiofrequency ablation — Radiofrequency ablation conducted per physicians' standard of care.
  Other Names: RFA

SUMMARY:
The purpose of this study is to evaluate pain the patient experienced following treatment of varicose veins with Varithena® compared to radiofrequency ablation.

DETAILED DESCRIPTION:
A study that evaluates pain following treatment of varicose veins in patients treated with Varithena® and those treated with RFA.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women; age 18 to 75 years
2. Bilateral incompetence of SFJ (reflux >1 second on duplex ultrasonography) associated with incompetence of the GSV in both legs
3. GSV diameter >5 mm measured from the superficial epigastric vein to 10 cm below the SFJ while in a standing position in both legs
4. Eligible to receive RFA treatment and Varithena® treatment
5. CEAP C2-C5 (inclusive)
6. Patient is participating in usual work and home activities with no changes anticipated for the duration of the study
7. Ability to comprehend and sign an informed consent and complete study questionnaires written in English
8. Ability to reliably use an electronic diary to record pain and analgesic/opioid use in accordance with the protocol

Exclusion Criteria:

1. Prior GSV treatment in either leg
2. Non-venous source of pain in either leg that could confound the results of the study
3. Use of chronic analgesic or opiate medications or medical history that could result in the regular use of pain medications during the study
4. History of deep vein thrombosis, pulmonary embolism or stroke, including evidence of prior or active DVT on duplex ultrasound
5. Deep venous reflux unless clinically insignificant in comparison to superficial reflux
6. Inability to wear post-procedure compression bandaging and stockings
7. Reduced mobility (unable to walk unaided for 5 minutes per waking hour)
8. Major surgery, prolonged hospitalization or pregnancy within 3 months of screening
9. Major co-existing disease (e.g., malignancy; pulmonary disease; renal or hepatic insufficiency; serious skin disease/condition that may compromise the ability of the patient to comply with the compression protocol, etc.)
10. Contraindications to Varithena® (e.g., acute thromboembolic disease) or RFA according to the manufacturer's prescribing information

    1. Varithena® contraindication due to known allergy to polidocanol
    2. RFA contraindication due to veins being too large
    3. RFA Contraindication due to veins being too tortuous
11. Known allergic response to polidocanol and/or multiple allergic reactions
12. Current or history of alcohol or drug abuse
13. Pregnant or lactating women
14. Women of childbearing potential not using effective contraception for at least one month prior to study treatment and/or unwilling to continue birth control for the duration of the study
15. Participation in a clinical study involving an investigational pharmaceutical product or device within the 3 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wright, MD, Study Director — BTG International Inc.
Locations (4):
- United States (4):
  - Coastal Vascular and Interventional, PLLC, Pensacola, Florida
  - Midwest Institute for Minimally Invasive Therapies, Melrose Park, Illinois
  - Venous Institute of Buffalo, Amherst, New York
  - Lake Washington Vascular, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Varithena® First Then Radiofrequency Ablation: Patients receive Varithena® treatment first in one leg, with 4-week follow-up period in Part 1; followed by Radiofrequency ablation in the other leg in Part 2.
  Varithena® treatment administered in accordance with full prescribing information and instructions for use.
  Radiofrequency ablation conducted per physicians' standard of care
- Radiofrequency Ablation First Than Varithena: Patients will receive radiofrequency ablation treatment first in one leg, with 4-week follow-up period in Part 1; followed by Varithena® in the other leg in Part 2.
  Varithena® treatment administered in accordance with full prescribing information and instructions for use.
  Radiofrequency ablation conducted per physicians' standard of care
Period: Part 1
Arm/Group | Varithena® First Then Radiofrequency Ablation | Radiofrequency Ablation First Than Varithena
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0
Period: Part 2
Arm/Group | Varithena® First Then Radiofrequency Ablation | Radiofrequency Ablation First Than Varithena
Started | 18 | 17
Completed | 17 | 16
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Varithena®: Varithena®: Varithena® treatment in accordance with full prescribing information and instructions for use followed by Radiofrequency ablation: Radiofrequency ablation conducted per physicians' standard of care.
  Radiofrequency ablation: Radiofrequency ablation conducted per physicians' standard of care followed by Varithena®: Varithena® treatment in accordance with full prescribing information and instructions for use
Arm/Group | Varithena®
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: 14-day average post-treatment pain using a VAS pain score. VAS pain score is an integer-valued, interval scale variable with range from 0 to 100 representing the spectrum from no pain to pain as bad as one can imagine.
Time Frame: 14 day average (0-100)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Varithena®: Varithena (polidocanol injectable foam) supplied as polidocanol solution 180 mg/18 mL (10 mg/mL) to be activated before use. Once activated, Varithena is a white injectable foam delivering a 1% polidocanol solution. Each milliliter of Varithena injectable foam contains 1.3 mg of polidocanol. Up to 5 mL per injection or 15 mL per treatment session could be used.
  Varithena®: Varithena® treatment in accordance with full prescribing information and instructions for use
  Radiofrequency ablation: Radiofrequency ablation conducted per physicians' standard of care.
- Radiofrequency Ablation: RFA procedures were conducted in accordance with the physician's standard of care and according to the manufacturer's instructions for use.
  Varithena®: Varithena® treatment in accordance with full prescribing information and instructions for use
  Radiofrequency ablation: Radiofrequency ablation conducted per physicians' standard of care.
Arm/Group | Varithena® | Radiofrequency Ablation
Number analyzed (Participants) | 33 | 33
units on a scale | 11.3 (2.90) | 9.5 (2.90)

2. Secondary Outcome: Procedural Pain
Description: degree of procedural pain perceived by the patient obtained immediately following the procedure using a VAS pain score. VAS pain score is an integer-valued, interval scale variable with range from 0 to 100 representing the spectrum from no pain to pain as bad as one can imagine
Time Frame: immediately following procedure
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Varithena®; Radiofrequency Ablation: Varithena® treatment in accordance with full prescribing information and instructions for use
  Radiofrequency ablation: Radiofrequency ablation conducted per physicians' standard of care.
Arm/Group | Varithena® | Radiofrequency Ablation
Number analyzed (Participants) | 33 | 33
units on a scale | 16.4 (3.53) | 17.8 (3.53)

3. Secondary Outcome: Patient Preference
Description: Patient preference for RFA or Varithena® using e-diary
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Varithena® | Radiofrequency Ablation
Number analyzed (Participants) | 33 | 33
Participants | 19 | 14

ADVERSE EVENTS:
Time Frame: A period of time ending at Week 4 (day 32)
Arm/Group | Varithena® | Radiofrequency Ablation
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 4/34 | 3/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varithena® (N=34) | Radiofrequency Ablation (N=34)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Phlebitis (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes